CLINICAL TRIAL: NCT00666107
Title: Pilot Study to Evaluate the Immunogenicity and Safety of the HPV Quadrivalent Vaccine (Gardasil) in HIV-infected Men
Brief Title: Pilot Study to Determine the Safety and Efficacy of Gardasil Against the Human Papilloma Virus (HPV) in HIV-infected Men
Acronym: MIRB #862
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: #33245
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2010-11

CONDITIONS: Anal Cancer; HIV Infections
Keywords: HPV; HIV; Gardasil; Vaccine
MeSH Terms: conditions — Anus Neoplasms; HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Gardasil — Intramuscular injections of Gardasil at Day 0, Month 2 and at Month 6
  Other Names: HPV quadrivalent vaccine

SUMMARY:
This study will investigate the efficacy and safety of the quadrivalent vaccine (Gardasil) against the human papilloma virus (HPV) in HIV (human immunodeficiency virus) infected males.

DETAILED DESCRIPTION:
This is a prospective pilot study that will attempt to enroll approximately 150-200 HIV-infected males followed regularly in the ID Primary Care Clinic at the VA Long Beach Healthcare System. All consenting patients will be given the HPV vaccine (Gardasil) in three intramuscular injections. Baseline antibody titers to HPV strains 16 and 18 will be obtained at day 0 and repeat levels will be obtained approximately 8 weeks after the completion of the vaccination series to determine whether patients without antibodies at baseline have now produced antibodies, or to determine the change in antibody levels in those patients who have evidence of antibodies prior to the first injection of the vaccine. Patients will undergo routine anal PAP smear with HPV DNA testing at baseline and another PAP smear/HPV test approximately 8 weeks after completion of the series. Patients will report any side effects of the vaccine to the PI. Patients will have blood work to monitor HIV-1 viral load and CD4 lymphocytes counts at various points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male veterans
* Age 18 or older
* HIV-positive
* Seen regularly in the ID Primary Care Clinic at the VA Long Beach Healthcare System

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Determine Geometric Mean Titers of anti-HPV 16 and anti-HPV 18 antibodies | nine months
Determine percentage of subjects who seroconverted or mounted a significant serologic response to each of the 2 antigens 16 and 18 | 8-9 months
Determine how many patients, if any, develop evidence of anal HPV infection, as measured by development of a positive HPV test. | 9 months
Determine if vaccinations will activate the subject's immune systems sufficiently that the HIV-1 viral load either increases from the baseline value, or becomes detectable and stays detectable after being undetectable at the baseline visit | nine months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Berman, M.D., Ph.D., Principal Investigator — Southern California Institute for Research and Education
Locations (1):
- VA Long Beach Healthcare System, Long Beach, California, United States

REFERENCES:
- [Background] Chin-Hong PV, Palefsky JM. Natural history and clinical management of anal human papillomavirus disease in men and women infected with human immunodeficiency virus. Clin Infect Dis. 2002 Nov 1;35(9):1127-34. doi: 10.1086/344057. Epub 2002 Oct 14. PMID 12384848
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Emeny RT, Wheeler CM, Jansen KU, Hunt WC, Fu TM, Smith JF, MacMullen S, Esser MT, Paliard X. Priming of human papillomavirus type 11-specific humoral and cellular immune responses in college-aged women with a virus-like particle vaccine. J Virol. 2002 Aug;76(15):7832-42. doi: 10.1128/jvi.76.15.7832-7842.2002. PMID 12097595
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Ault KA, Giuliano AR, Wheeler CM, Koutsky LA, Malm C, Lehtinen M, Skjeldestad FE, Olsson SE, Steinwall M, Brown DR, Kurman RJ, Ronnett BM, Stoler MH, Ferenczy A, Harper DM, Tamms GM, Yu J, Lupinacci L, Railkar R, Taddeo FJ, Jansen KU, Esser MT, Sings HL, Saah AJ, Barr E. Prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in young women: a randomised double-blind placebo-controlled multicentre phase II efficacy trial. Lancet Oncol. 2005 May;6(5):271-8. doi: 10.1016/S1470-2045(05)70101-7. PMID 15863374
- [Background] Olsson SE, Villa LL, Costa RL, Petta CA, Andrade RP, Malm C, Iversen OE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, von Krogh G, Lehtinen M, Paavonen J, Tamms GM, Giacoletti K, Lupinacci L, Esser MT, Vuocolo SC, Saah AJ, Barr E. Induction of immune memory following administration of a prophylactic quadrivalent human papillomavirus (HPV) types 6/11/16/18 L1 virus-like particle (VLP) vaccine. Vaccine. 2007 Jun 21;25(26):4931-9. doi: 10.1016/j.vaccine.2007.03.049. Epub 2007 Apr 20. PMID 17499406
- [Background] Bower M, Powles T, Newsom-Davis T, Thirlwell C, Stebbing J, Mandalia S, Nelson M, Gazzard B. HIV-associated anal cancer: has highly active antiretroviral therapy reduced the incidence or improved the outcome? J Acquir Immune Defic Syndr. 2004 Dec 15;37(5):1563-5. doi: 10.1097/00126334-200412150-00004. PMID 15577408
- [Background] Bozzette SA, Phillips B, Asch S, Gifford AL, Lenert L, Menke T, Ortiz E, Owens D, Deyton L. Quality Enhancement Research Initiative for human immunodeficiency virus/acquired immunodeficiency syndrome: framework and plan. HIV-QUERI Executive Committee. Med Care. 2000 Jun;38(6 Suppl 1):I60-9. doi: 10.1097/00005650-200006001-00007. PMID 10843271